#### The GlaxoSmithKline group of companies

| Division | : | Worldwide Development |
|------------------|---|-----------------------------------|
| Information Type | : | Reporting and Analysis Plan (RAP) |

| Title | : | Reporting and Analysis Plan for 204678 |
|---|---|---|
| | | A single centre, open-label, parallel-group, single oral dose<br>study to evaluate the pharmacokinetic, safety and tolerability<br>of Pyrimethamine in healthy Japanese and Caucasian male<br>subjects |
| <b>Compound Number</b> | : | GR99352 |
| Effective Date | : | 15-SEP-2017 |

# **Description:**

- The purpose of this RAP is to describe the planned analyses and output to be included in the Clinical Study Report for Protocol 204678.
- This RAP is intended to describe the Pharmacokinetic (PK) and safety analyses required for the study.
- This RAP will be provided to the study team members to convey the content of the Statistical Analysis Complete (SAC) deliverable.

#### Author's Name and Functional Area:

| PPD | 23-AUG-2017 |
|---|---|
| Biostatistics Group 1, Biomedical Data Sciences Dept. | 20 110 0 2017 |
| Clinical Pharmacology & Science Promotion Office. | 23-AUG-2017 |
| Statistical Programming & Reporting Group, Biomedical Data Sciences Dept. | 23-AUG-2017 |

#### Approved by (Approvals captured electronically in CARS system):

| PPD | | |
|---|---|---|
| Manager, Stat | istical Programming & Reporting Group, Biomedical | 15-SEP-2017 |
| Data Sciences | Dept. | |
| PPD | | 15 GED 2015 |
| Manager, Biostatistics Group 1, Biomedical Data Sciences Dept. 15-SEP-2017 | | |

Copyright 2017 the GlaxoSmithKline group of companies. All rights reserved. Unauthorised copying or use of this information is prohibited.

# **TABLE OF CONTENTS**

| | | | PAGE |
|---|---|---|---|
| 1. | REPO | RTING & ANALYSIS PLAN SYNPOSIS | 4 |
| | 1.1. | History | |
| 2. | SLIMA | MARY OF KEY PROTOCOL INFORMATION | 6 |
| ۷. | 2.1. | Changes to the Protocol Defined Statistical Analysis Plan | |
| | 2.2. | Study Objective(s) and Endpoint(s) | |
| | 2.3. | Study Design | |
| | 2.4. | Statistical Hypotheses | |
| 3. | PI ANI | NED ANALYSES | 7 |
| Ο. | 3.1. | Interim Analyses | |
| | 3.2. | Final Analyses | |
| 4. | ANAI ` | YSIS POPULATIONS | 8 |
| | 4.1. | Protocol Deviations | |
| 5. | | SIDERATIONS FOR DATA ANALYSES AND DATA HANDLING | |
| | CONV | 'ENTIONS | 9 |
| 6. | STUD | Y POPULATION ANALYSES | 10 |
| | 6.1. | Overview of Planned Analyses | 10 |
| 7. | SAFE | TY ANALYSES | 11 |
| | 7.1. | Overview of Planned Analyses | |
| | 7.2. | Overview of Planned Clinical Laboratory Analyses | |
| | 7.3. | Overview of Planned Other Safety Analyses | 12 |
| 8. | PHAR | MACOKINETIC ANALYSES | 13 |
| | 8.1. | Overview of Planned Pharmacokinetic Analyses | 13 |
| | 8.2. | Drug Concentration Measures | |
| | 8.3. | Pharmacokinetic Parameters | |
| | | 8.3.1. Derived Pharmacokinetic Parameters | |
| | | 8.3.2. Summary of Pharmacokinetic Parameters | 16 |
| 9. | REFE | RENCES | 17 |
| 10 | ∧ DDE | NDICES | 10 |
| 10. | 10.1. | Appendix 1: Protocol Deviation Management | |
| | 10.1. | Appendix 2: Time & Events | |
| | 10.2. | 10.2.1. Protocol Defined Time & Event | |
| | 10.3. | Appendix 3: Treatment States and Phases | |
| | 10101 | 10.3.1. Treatment Phases | |
| | 10.4. | Appendix 4: Data Display Standards & Handling Conventions | |
| | | 10.4.1. Study Treatment & Sub-group Display Descriptors | |
| | | 10.4.2. Baseline Definition & Derivations | |
| | | 10.4.3. Reporting Process & Standards | |
| | 10.5. | Appendix 5: Derived and Transformed Data | |
| | | 10.5.1. General | |
| | | 10.5.2. Study Population | 26 |

#### CONFIDENTIAL

| | 10.5.3. | Safety | 27 |
|---|---|---|---|
| | 10.5.4. | · | |
| 10.6. | <b>Appendix</b> | 6: Premature Withdrawals & Handling of Missing Data | 29 |
| | | Premature Withdrawals | |
| | 10.6.2. | Handling of Missing Data | 29 |
| 10.7. | <b>Appendix</b> | 7: Values of Potential Clinical Importance | |
| | 10.7.1. | Laboratory Values | 30 |
| | 10.7.2. | | |
| | 10.7.3. | Vital Signs | 31 |
| 10.8. | <b>Appendix</b> | 8 – Abbreviations & Trade Marks | 32 |
| | 10.8.1. | Abbreviations | 32 |
| | 10.8.2. | Trademarks | 32 |
| 10.9. | <b>Appendix</b> | 9: List of Data Displays | 33 |
| | 10.9.1. | Data Display Numbering | 33 |
| | 10.9.2. | Mock Example Shell Referencing | 33 |
| | 10.9.3. | Deliverable [Priority] | |
| | 10.9.4. | Study Population Tables | 34 |
| | 10.9.5. | Safety Tables | 35 |
| | 10.9.6. | Pharmacokinetic Tables | 37 |
| | 10.9.7. | Pharmacokinetic Figures | 38 |
| | 10.9.8. | ICH Listings | 40 |
| 10.10. | <b>Appendix</b> | 10: Example Mock Shells for Data Displays | 43 |

# 1. REPORTING & ANALYSIS PLAN SYNPOSIS

| Overview | Key Elements of the RAP |
|---|---|
| Purpose | The purpose of this RAP is to describe the planned analyses and output to be included in the Clinical Study Report for Protocol 204678. |
| Protocol | • This RAP is based on the original protocol Dated:19/JUL/2017 of study204678 (GSK Document Number.: 2017N318316_00). |
| Primary<br>Objective | • To investigate PK following a single oral dose of Pyrimethamine 50 mg in fasted healthy Japanese male subjects. |
| Primary<br>Endpoint | • Cmax, AUC(0-t), AUC(0-inf), AUC(0-24), tmax, t1/2, CL/F, Vd/F from the plasma concentrations of Pyrimethamine in healthy Japanese male subjects, as data permit. |
| Study Design | This study will be a single centre, open-label, parallel-group, single oral dose study to evaluate the pharmacokinetic (PK), safety and tolerability of Pyrimethamine in healthy Japanese and Caucasian male subjects. |
| | • Sufficient Japanese and Caucasian healthy male volunteer subjects will be enrolled such that 6 subjects of each population complete dosing and critical assessments. |
| Analysis<br>Populations | Screened: Consisting of all participants screened in the study. |
| | • Screening Failure: Participants who sign the ICF in the study but are never subsequently administered study treatment. |
| | Safety: All participants who take at least one dose of study treatment. |
| | Pharmacokinetic: This population is defined as all participants administered at least one dose of study treatment and who have PK sample taken and analyzed. |
| Hypothesis | • The objectives of this study are to evaluate safety and tolerability of Pyrimethamine and to estimate Pyrimethamine pharmacokinetic parameters in healthy male Japanese and Caucasian subjects. No formal statistical hypotheses will be tested. Descriptive statistics will be used to assess safety and tolerability objectives. An estimation approach will be used to address the pharmacokinetic study objectives, where point estimates and corresponding 95% confidence intervals will be constructed, unless otherwise stated. |

| Overview | Key Elements of the RAP |
|---|---|
| Pharmacokinetic<br>Analyses | • Individual Pyrimethamine plasma concentration-time profiles (by group, and subject) and median/mean (±SD) profiles by group will be plotted and listed. |
| | • Plasma concentration time data for Pyrimethamine will be analyzed by non-compartmental methods using Phoenix WinNonlin (version 6.3 or higher) and all derived PK parameters will be graphically presented, summarised and listed. No formal statistical analyses will be conducted. |
| Safety Analyses | Safety data will be presented in tabular and/or graphical format and summarised descriptively. |

# 1.1. History

| Version | Issue Date | Amendments | Reason |
|---------|-------------|-------------------------|--------|
| 00 | 15-SEP-2017 | Original (New document) | - |

# 2. SUMMARY OF KEY PROTOCOL INFORMATION

# 2.1. Changes to the Protocol Defined Statistical Analysis Plan

There were no changes or deviations to the originally planned statistical analysis specified in the protocol (Dated: 19/JUL/2017).

# 2.2. Study Objective(s) and Endpoint(s)

| Objectives | Endpoints |
|---|---|
| Primary Objectives | Primary Endpoints |
| To investigate PK following single<br>dose of Pyrimethamine 50 mg in<br>fasted status in healthy Japanese<br>male subjects. | Cmax, AUC(0-t), AUC(0-inf), AUC(0-24), tmax, t1/2, CL/F, Vd/F of the plasma concentration of Pyrimethamine in healthy Japanese male subjects, as data permit. |
| Secondary Objectives | Secondary Endpoint |
| To investigate PK following single<br>dose of Pyrimethamine 50 mg in<br>fasted status in healthy Caucasian<br>male subjects. | Cmax, AUC(0-t), AUC(0-inf), AUC(0-24), tmax, t1/2, CL/F, Vd/F of the plasma concentration of Pyrimethamine in healthy Caucasian male subjects, as data permit. |
| To assess safety and tolerability<br>following single dose of<br>Pyrimethamine in fasted status in<br>healthy Japanese and Caucasian<br>male subjects. | AE and change from the baseline of clinical laboratory values, vital signs and ECG. |

## 2.3. Study Design

| Overview of S | Overview of Study Design and Key Features |
|---|---|
| Design<br>Features | |
| Dosing | <ul> <li>Subjects will have a screening visit within 30 days prior to the first dose of study treatment, one treatment period, and re-visits 15 (±1) and 22 (±1) days after the dose for follow-up assessments including PK sampling.</li> <li>Subjects will be housed in the Clinical Research Unit from Day -1 through Day 8, and return to the unit on Day 15 (±1) and 22 (±1) for the remaining PK samples and safety assessments post dose.</li> <li>During the treatment period, subjects will receive single dose of Pyrimethamine 50 mg in the fasted state after overnight fast (at least 10 hours). Calcium folinate 15 mg will be coadministered with Pyrimethamine at Day 1, and will continue to be administered once a day until Day 8.</li> <li>Blood sampling for PK analysis and safety assessments will be performed prior to dosing and over 22 days after dosing. The duration of each subject's participation will be approximately 2 months from screening to the follow-up.</li> </ul> |
| Treatment<br>Assignment | <ul> <li>Sufficient Japanese and Caucasian healthy male subjects will be enrolled<br/>such that 6 subjects of each population complete dosing and critical<br/>assessments.</li> </ul> |
| Interim<br>Analysis | No interim analyses will be planned. |

# 2.4. Statistical Hypotheses

The objectives of this study are to evaluate safety and tolerability of Pyrimethamine and to estimate Pyrimethamine pharmacokinetic parameters in healthy Japanese and Caucasian male subjects. No formal statistical hypotheses will be tested. Descriptive statistics will be used to assess safety and tolerability objectives by group (Japanese, Caucasian). An estimation approach will be used to address the pharmacokinetic study objectives, where point estimates and corresponding 95% confidence intervals will be constructed, unless otherwise stated.

# 3. PLANNED ANALYSES

# 3.1. Interim Analyses

An interim analysis is not planned.

# 3.2. Final Analyses

The final planned primary analyses will be performed after the completion of the following sequential steps:

- 1. All subjects have completed the study as defined in the protocol.
- 2. All required database cleaning activities have been completed and final database release and database freeze has been declared by Data Management.
- 3. Even though single arm study, randomisation codes have been distributed according to RandAll NG procedures.

#### 4. ANALYSIS POPULATIONS

| Population | Definition / Criteria | Analyses Evaluated |
|---|---|---|
| Screened | Consisting of all participants screened in the study | Study Population |
| Screening Failure | Participants who sign the ICF in the study but are never subsequently administered study treatment. All participants who sign the ICF have the screening test in the study. | Study Population |
| Safety | All participants who take at least one dose of study treatment. | <ul><li>Study Population</li><li>Safety</li></ul> |
| Pharmacokinetic | This population is defined as all participants administered at least one dose of study treatment and who have PK sample taken and analysed. | • PK |

#### 4.1. Protocol Deviations

- Important protocol deviations (including deviations related to study inclusion/exclusion criteria, conduct of the trial, patient management or patient assessment) will be summarised and listed.
- Protocol deviations will be tracked by the study team throughout the conduct of the study in accordance with the Protocol Deviation Management Plan.
  - Data will be reviewed prior to freezing the database to ensure all important deviations and deviations which may lead to exclusion from the analysis are captured and categorised on the protocol deviations dataset.
  - This dataset will be the basis for the summaries and listings of protocol deviations.
- A separate listing of all inclusion/exclusion criteria deviations will also be provided. This will be based on data as recorded on the inclusion/exclusion page of the eCRF.

# 5. CONSIDERATIONS FOR DATA ANALYSES AND DATA HANDLING CONVENTIONS

Table 1 provides an overview of appendices within the RAP for outlining general considerations for data analyses and data handling conventions.

Table 1 Overview of Appendices

| Section | Component |
|---------|--------------------------------------------------------------|
| 10.1 | Appendix 1: Protocol Deviation Management |
| 10.2 | Appendix 2: Time & Events |
| 10.3 | Appendix 3: Treatment States and Phases |
| 10.4 | Appendix 4: Data Display Standards & Handling Conventions |
| 10.5 | Appendix 5: Derived and Transformed Data |
| 10.6 | Appendix 6: Premature Withdrawals & Handling of Missing Data |
| 10.7 | Appendix 7: Values of Potential Clinical Importance |

## 6. STUDY POPULATION ANALYSES

# 6.1. Overview of Planned Analyses

The study population analyses will be based on the Safety population, unless otherwise specified.

Table 2 provides an overview of the planned study population analyses, with full details of data displays being presented in Appendix 9: List of Data Displays.

 Table 2
 Overview of Planned Study Population Analyses

| Display Type | Data | Displays Gene | rated |
|---|---|---|---|
| | Table | Figure | Listing |
| Subject Disposition | | | |
| Subject Disposition and Reason for Study Withdrawal | Υ | | Υ |
| Screening Status and Reasons for Screen Failure | Y | | Υ |
| Protocol Deviations | | | |
| Important Protocol Deviations | Υ | | Υ |
| Subjects with Inclusion/Exclusion Criteria Deviations | | | Υ |
| Populations Analysed | | | |
| Study Populations | Y | | |
| Subjects Excluded from Any Population | | | Υ |
| Demographic and Baseline Characteristics | | | |
| Demographic Characteristics | Υ | | Υ |
| Demographic Characteristics for Screening Failure | | | Υ |
| Age Ranges | Y | | |
| Race and Racial Combinations | Y | | Υ |
| Race and Racal Combination for Failure | | | Υ |
| Medical Conditions and Concomitant Medications | | | |
| Medical Conditions | | | Υ |
| Concomitant Medications | | | Y |
| Exposure and Treatment Compliance | | | |
| Exposure to Study Treatment | | | Υ |

#### NOTES:

• Y = Yes display generated.

# 7. SAFETY ANALYSES

The safety analyses will be based on the Safety population, unless otherwise specified.

# 7.1. Overview of Planned Analyses

Table 3 provides an overview of the planned analyses, with further details of data displays being presented in Appendix 9: List of Data Displays.

Table 3 Overview of Planned Safety Analyses

| Display Type | | Absolute | |
|---|---|---|---|
| | Sur | nmary | Individual |
| | Т | F | L |
| Adverse Events (AEs) | | | |
| All AEs by SOC and PT | Υ | | Υ |
| All AEs by Maximum Intensity | Υ | | |
| Drug-Related AEs by SOC and PT | Υ | | |
| Drug-Related AEs by Maximum Intensity | Υ | | |
| Subject Numbers for Individual AEs | | | Υ |
| Relationship Between AE SOCs, PT and Verbatim Text | | | Υ |
| Serious and Other Significant AEs | | | |
| Serious AEs | | | Υ |
| AEs Leading to Withdrawal from Study | | | Υ |

#### NOTES:

- T = Table, F = Figures, L = Listings, Y = Yes display generated, SOC = System Organ Class, PT = Preferred Term.
- Summary = Represents TF related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.

## 7.2. Overview of Planned Clinical Laboratory Analyses

Table 4 provides an overview of the planned analyses, with further details of data displays being presented in Appendix 9: List of Data Displays.

Table 4 Overview of Planned Clinical Laboratory Analyses

| Display Type | | Abs | olute | Change from BL | | |
|---|---|---|---|---|---|---|
| | Sum | Summary Individual | | Sumr | nary | Individual |
| | Т | F | L | Т | F | L |
| Chemistry | | • | | | • | |
| Chemistry Data | Υ | | Υ | Υ | | Υ |
| Chemistry Results Relative to Normal Range | | | | Υ | | |
| All Chemistry Data for Subjects with any Value of Potential Clinical Concern/PCI | | | Y | | | |

| Display Type | | Abs | olute | Change from BL | | |
|---|---|---|---|---|---|---|
| | Sum | mary | Individual | Sumr | nary | Individual |
| | Т | F | L | Т | F | L |
| Hematology | | | | | | |
| Hematology Data | Υ | | Υ | Υ | | Υ |
| Hematology Results Relative to Normal Range | | | | Υ | | |
| All Hematology Data for Subjects with any Value of Potential Clinical Concern/PCI | | | Y | | | |
| Urinalysis | | | | | | |
| Dipstick Data (Glucose, Protein, Blood, Ketones, Bilirubin, Urobilinogen) | Υ | | Y* | | | |
| Gravity and pH | Υ | | Υ | | | |
| Hepatobiliary (Liver) | | | | | | |
| Liver Monitoring/Stopping Event Reporting | | | Υ | | | |
| Medical Conditions for Subjects with Liver Stopping Events | | | Y | | | |
| Substance Use for Subjects with Liver Stopping Events | | | Y | | | |

#### NOTES:

- T = Table, F = Figures, L = Listings, Y = Yes display generated, PCI = Potential Clinical Importance
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
   Individual = Represents FL related to any displays of individual subject observed raw data.

# 7.3. Overview of Planned Other Safety Analyses

Table 5 provides an overview of the planned analyses, with further details of data displays being presented in Appendix 9: List of Data Displays.

Table 5 Overview of Planned Other Safety Analyses

| Display Type | | Abs | olute | Change from BL | | |
|---|---|---|---|---|---|---|
| | Sum | mary | Individual | Sumn | nary | Individual |
| | Т | F | L | T | F | L |
| ECG | | | | | | |
| ECG Findings | Υ | | Υ | | | |
| ECG Values | Υ | | Υ | Υ | | Y |
| All ECG Values for Subjects with any Value of PCI | | | Υ | | | |
| Vital Signs | | | | | | |
| Vitals Values | Υ | | Υ | Υ | | Υ |
| All Vital Signs for Subjects with any Value of PCI | | | Υ | | | |

#### NOTES:

- T = Table, F = Figures, L = Listings, Y = Yes display generated, PCI = Potential Clinical Importance
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.

<sup>\*:</sup> If blood or protein is abnormal, microscopic examination will be included.

#### 8. PHARMACOKINETIC ANALYSES

## 8.1. Overview of Planned Pharmacokinetic Analyses

The pharmacokinetic (PK) analyses will be based on the Pharmacokinetic population, unless otherwise specified.

Table 6 provides an overview of the planned analyses, with full details being presented in Appendix 9: List of Data Displays.

Table 6 Overview of Planned Pharmacokinetic Analyses

| Display Type | | Untrans | formed | | | Log-Trar | nsformed | |
|---|---|---|---|---|---|---|---|---|
| | Summary | | Individual | | Summary | | Individual | |
| | F | T | F | L | F | T | F | L |
| Plasma Drug Concentrations | Υ [1] [2] | Υ | Υ [1] | Υ | | | | |
| Derived PK Parameters | Υ | Υ | | Υ | | Υ | | |

#### NOTES:

- T = Table, F = Figures, L = Listings, Y = Yes display generated.
- Summary = Represents TFL related to any summaries (descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.
- 1. Linear and Semi-Log plots will be created on the same display.
- 2. Separate Mean (± SD) and Median plots will be generated.

# 8.2. Drug Concentration Measures

Plasma concentrations of Pyrimethamine at each nominal time will be listed and summarised by group. Standard summary statistics will be calculated (i.e. mean, standard deviation, median, minimum and maximum).

Individual plasma concentration-time profiles and median/mean profiles by group will be plotted. Each of the figures will contain one plot on the untransformed scale (i.e. a linear plot) and one plot on the log transformed scale (i.e. log-linear plot).

All individual plasma concentration-time profiles will be plotted. Each of the figures will contain one plot on the untransformed scale (i.e. a linear plot) and one plot on the log transformed scale (i.e. log-linear plot).

Refer to Appendix 4: Data Display Standards & Handling Conventions (Section 10.4.3 Reporting Process & Standards).

#### 8.3. Pharmacokinetic Parameters

#### 8.3.1. Derived Pharmacokinetic Parameters

- Derivation of pharmacokinetic parameters will be performed by, or under the direct auspices of, Clinical Pharmacology & Science Promotion Office, GlaxoSmithKline K.K.
- Refer to Appendix 4: Data Display Standards & Handling Conventions (Section 10.4.3 Reporting Process & Standards).
- The pharmacokinetic parameters will be calculated by non-compartmental analysis using Phoenix WinNonlin (version 6.3 or higher)
- All calculations of non-compartmental parameters will be based on actual sampling times recorded during the study.

Pharmacokinetic parameters described in Table 7 will be determined from plasma Pyrimethamine concentration-time data, as data permits.

# Table 7 Derived Pharmacokinetic Parameters

| Parameter | Parameter Description |
|---|---|
| AUC(0-24) | Area under the concentration-time curve will be calculated to fixed nominal time 24 hours after administration (AUC(0-24)), using the combination of linear and logarithmic trapezoidal methods (i.e., Linear Up/Log Down calculation method in Phoenix WinNonlin). If a sampling time deviation occurred at nominal time 24 hours after administration (and 24 < t), AUC(0-24) will be calculated using the concentration at time 24 hours after administration post-dose estimated by the method of interpolation. If nominal time 24 hours after administration > t (or if the concentration at time 24 hours after administration was below the limit of quantification), then the concentration (y) at time 24 hours after administration is estimated using $\lambda z$ and last observed Ct according to the formula: $y = Ct(obser) \times e^{-lambda_z z(24-t)}$ Then the following equation will be used to calculate AUC(0-24) where t is the time of last quantifiable plasma concentration. $AUC(0-24) = AUC(0-t) + AUC(t-24)$ |
| AUC(0-t) | If lambda_z is not estimable, AUC(0-24) is not calculated (when 24 > t). Area under the concentration-time curve from time zero time (pre-dose) to the time of last quantifiable concentration (AUC(0-t)) will be calculated by a combination of linear and logarithmic trapezoidal methods. The linear trapezoidal method will be employed for all incremental trapezoids arising from increasing concentrations and the logarithmic trapezoidal method will be used for those arising from decreasing concentrations (i.e., Linear Up/Log Down calculation method in Phoenix WinNonlinl). |
| AUC(0-inf) | Area under the concentration-time curve from zero time (pre-dose) extrapolated to infinite time (AUC(0-inf)) will be calculated as follows: AUC(0-inf) = AUC(0-t) + C(t) / lambda_z |
| %AUCex | The percentage of AUC (0-∞) obtained by extrapolation (%AUCex) will be calculated as: %AUCex = [AUC(0-inf) – AUC(0-t)] / AUC(0-inf) x 100 |
| Cmax | Maximum observed concentration will be obtained directly from the concentration-time data. |
| Tmax | Time to first occurrence of Cmax will be obtained directly from the concentration-time data. |
| t½ | Apparent terminal phase half-life will be calculated as: t½ = In2 / lambda_z |
| Tlast | The time of the last measurable (positive) concentration. |
| lambda_z | The first order rate constant associated with the terminal (log-linear) portion of the curve. |
| lambda_z<br>lower | The lower limit on time for values to be included in the calculation of lambda_z. |
| lambda_z<br>upper | The upper limit on time for values to be included in the calculation of lambda_z. |
| #pts | The number of time points used in computing lambda_z. |
| R-square | Square of the correlation coefficient. |
| CL/F | Apparent clearance following oral dosing will be calculated as: CL/F = Dose / AUC (0-inf) |
| Vd/F | Apparent volume of distribution following oral dosing will be calculated as: Vd/F = Dose / lambda_z * AUC(0-inf) |

#### NOTES:

- Additional parameters may be included as required.
- Lambda\_z is the terminal phase rate constant.
- Ct is the last observed quantifiable concentration.

## 8.3.2. Summary of Pharmacokinetic Parameters

- For each of these parameters, except for tmax, the following summary statistics will be calculated for each treatment:
  - o Non-transformed: median, maximum, minimum, arithmetic mean, 95% confidence interval for the arithmetic mean and standard deviation
  - Loge-transformed: geometric mean, 95% confidence interval for the geometric mean, standard deviation of logarithmically transformed data and between geometric coefficient of variation (CVb (%))
- For tmax, median, maximum, minimum, arithmetic mean, standard deviation and 95% Confidence Interval (CI) for the arithmetic mean will be calculated.
- An exploratory analysis will be performed using PK parameter plots in order to assess the results in Japanese and Caucasian subjects. Plots of AUC(0-t), AUC(0-inf), Cmax and T1/2 versus group (Japanese, Caucasian) will be produced.

# 9. REFERENCES

GlaxoSmithKline Document Numbers 2017N318316\_00 Study Protocol of 204678. A single centre, open-label, parallel, single oral dose study to evaluate the pharmacokinetic, safety and tolerability of Pyrimethamine in healthy Japanese and Caucasian subjects (Effective date: 19-JUL-17)

# 10. APPENDICES

| Section | Appendix |
|---|---|
| RAP Section 4 | : Analysis Populations |
| Section 10.1 | Appendix 1: Protocol Deviation Management |
| RAP Section 5 | : General Considerations for Data Analyses & Data Handling Conventions |
| Section 10.2 | Appendix 2: Time and Events |
| Section 10.3 | Appendix 3: Treatment States & Phases |
| Section 10.4 | Appendix 4: Data Display Standards & Handling Conventions |
| | Study Treatment & Sub-group Display Descriptors |
| | Baseline Definitions & Derivations |
| | Reporting Process & Standards |
| Section 10.5 | Appendix 5: Derived and Transformed Data |
| | General |
| | Study Population |
| | Safety |
| | Pharmacokinetic |
| Section 10.6 | Appendix 6: Premature Withdrawals & Handling of Missing Data |
| | General |
| | Study Population & Safety |
| Section 10.7 | Appendix 7: Values of Potential Clinical Importance |
| | Laboratory Values |
| | • ECG |
| | Vital Signs |
| Other RAP App | endices |
| Section 10.8 | Appendix 8: Abbreviations & Trade Marks |
| Section 10.9 | Appendix 9: List of Data Displays |
| Section 10.10 | Appendix 10: Example Mock Shells for Data Displays |

# 10.1. Appendix 1: Protocol Deviation Management

Details will be referred latest Protocol Deviation Management Plan and data handling will be decided prior to final data base release.

# 10.2. Appendix 2: Time & Events

# 10.2.1. Protocol Defined Time & Event

| | Scr | Day<br>-1 | | | | Day 1 | | | | Day<br>2 | Day<br>3 | Day<br>4 | Day<br>5 | Day<br>6 | Day<br>7 | Day<br>8 | Day<br>15 <sup>4</sup> | Follow-<br>up<br>Day 22 <sup>4</sup> |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | -' | Pre | 0 h | 1 h | 2 h | 4 h | 6 h | 12 h | 24 h | 48 h | 72 h | 96 h | 120<br>h | 144<br>h | 168<br>h | 336<br>h | 504 h |
| Admission to Unit | | Χ | | | | | | | | | | | | | | | | |
| Informed consent | Х | | | | | | | | | | | | | | | | | |
| Subject<br>demography/Medical<br>history | Х | | | | | | | | | | | | | | | | | |
| Physical examination | Х | Χ | | | | | | | | Х | Χ | Χ | Χ | Χ | Χ | Χ | | Χ |
| 12-lead ECG | Х | | Χ | | | | Χ | | Х | Х | Χ | | | | | | | Χ |
| Vital signs | Х | | Χ | | | | Х | | Х | Х | Х | Х | Х | Х | Χ | Χ | Χ | Χ |
| Urine drug screen | Х | Χ | | | | | | | | | | | | | | | | |
| Alcohol breath test | Х | Χ | | | | | | | | | | | | | | | | |
| CO breath test | Х | Χ | | | | | | | | | | | | | | | | |
| Serological test | Х | | | | | | | | | | | | | | | | | |
| Haematology, clinical chemistry and urinalysis | Х | Х | | | | | | | | Х | | | Х | | | Χ | Х | Х |
| Study treatment dosing | | | | Х | | | | | | | | | | | | | | |
| Calcium folinate dosing | | | | X 1 | | | | | | Х | Х | Х | Х | Х | Χ | Χ | | |
| PK Sampling | | | Χ | | Х | Х | Х | Х | Х | Х | Х | Х | | Х | | Χ | Χ | Χ |
| SAEs <sup>2</sup> | ←===================================== | | | | | | | | | | | | | | | | | |
| AEs <sup>3</sup> | | | | <b>←===</b> | | | | | | | | | | | | | | ====→ |
| Con Med review | <b>←==</b> : | ===== | ===== | ====== | | ===== | | | ===== | | | | ===== | | | | ===== | ====> |
| Discharge | | | | | | | | | | | | | | | | Χ | | |
| Outpatient Visit | Х | | | | | | | | | | | | | | | | Χ | Χ |

#### **CONFIDENTIAL**

204678

- Calcium folinate will be coadministered with Pyrimethamine on Day 1.
   All SAEs will be collected from the signing of the ICF until the follow-up visit at the time points specified.
- All AEs will be collected from the start of treatment until the follow-up visit at the time points specified.
   Subjects will return to the unit on Day 15 (±1) and 22 (±1) for the remaining PK samples and safety assessments post dose.

# 10.3. Appendix 3: Treatment States and Phases

#### 10.3.1. Treatment Phases

Assessments and events will be classified according to the time of occurrence relative to the assessment date.

# 10.3.1.1. Treatment States for AE Data

| Treatment State | Definition |
|---|---|
| Pre-Treatment | AE Start Date < Study Treatment Start Date and Time |
| On treatment | Dosing Start Date and Time in each group ≤ AE Start Date and Time |
| Onset Time Since<br>First Dose | If Dosing Start Date and Time > AE Onset Date and Time = AE Onset Date and Time − Dosing Start Date and Time If dosing Start Date and Time ≤ AE Onset Date and Time = AE Onset Date and Time - |
| (Minute) | Dosing Start Date and Time +1 Missing otherwise |
| Onset Time Since<br>Last Dose<br>(Minute) | AE Start Date and Time – Most Recent Treatment Start Date and Time + 1 |
| Duration (Minute) | AE Resolution Date and Time – AE Onset Date and Time + 1 |
| Drug-related | If relationship is marked 'YES' on eCRF |

# 10.4. Appendix 4: Data Display Standards & Handling Conventions

#### 10.4.1. Study Treatment & Sub-group Display Descriptors

| Treatment Group Descriptions | | | |
|---|---|---|---|
| RandAll NG Data Displays for Reporting | | | |
| Schedule | Description | Description | Order [1] |
| 1 | D | Caucasian | 2 |
| 2 | D | Japanese | 1 |

#### NOTES:

#### 10.4.2. Baseline Definition & Derivations

#### 10.4.2.1. Baseline Definitions

| Parameter | Study Assessments Considered As Baseline | | | Baseline Used in |
|---|---|---|---|---|
| Faiailletei | Screening | Day -1 | Day 1<br>(Pre-Dose) | Data Display |
| Safety | | | | |
| 12 Lead ECG & Vital Signs | Х | | Х | Day 1<br>(Pre Dose) |
| Haematology | Х | Х | | Day -1 |
| Clinical Chemistry | X | Χ | | Day -1 |

#### 10.4.2.2. Derivations and Handling of Missing Baseline Data

| Definition | Reporting Details |
|----------------------|------------------------------------|
| Change from Baseline | = Post-Dose Visit Value – Baseline |

#### NOTES:

- Unless otherwise specified, the baseline definitions specified in Section 10.4.2.1 Baseline Definitions will be used for derivations for endpoints / parameters and indicated on summaries and listings.
- Unless otherwise stated, if baseline data is missing no derivation will be performed and will be set to missing.

# 10.4.3. Reporting Process & Standards

| Reporting Area | |
|----------------------------------------------------------------|-----|
| Software | |
| The currently supported versions of SAS software will be used. | |
| Reporting Area | |
| HARP Server | N/A |

<sup>1.</sup> Order represents treatments being presented in TFL, as appropriate.

| Reporting Area | |
|----------------|-----|
| HARP Area | N/A |
| QC Spreadsheet | N/A |

#### **Analysis Datasets**

 Analysis datasets will be created according to CDISC standards (SDTM IG Version 3.1.3 & AdaM IG Version 1.0).

#### **Generation of RTF Files**

N/A

#### **Reporting Standards**

#### General

- The current GSK Integrated Data Standards Library (IDSL) will be applied for reporting, unless otherwise stated:
  - 4.03 to 4.23: General Principles
  - 5.01 to 5.08: Principles Related to Data Listings
  - 6.01 to 6.11: Principles Related to Summary Tables
  - 7.01 to 7.13: Principles Related to Graphics

#### **Formats**

- All data will be reported according to the actual treatment the subject received unless otherwise stated.
- GSK IDSL Statistical Principles (4.24) for decimal places (DP's) will be adopted for reporting of data based on the raw data collected.
- Numeric data will be reported at the precision collected on the eCRF.
  - The reported precision from non eCRF sources will follow the IDSL statistical principles but may be adjusted to a clinically interpretable number of DP's.

#### Planned and Actual Time

- Reporting for tables, figures and formal statistical analyses :
  - Planned time relative to dosing will be used in figures, summaries, statistical analyses and calculation of any derived parameters, unless otherwise stated..
  - For PK parameters derivation, actual times are used.
  - The impact of any major deviation from the planned assessment times and/or scheduled visit days on the analyses and interpretation of the results will be assessed as appropriate.
- Reporting for Data Listings:
  - Planned and actual time relative to study drug dosing will be shown in listings (Refer to IDSL Statistical Principle 5.05.1).
  - Unscheduled or unplanned readings will be presented within the subject's listings.
  - Visits outside the protocol defined time-windows (i.e. recorded as protocol deviations) will be included in listings but omitted from figures, summaries and statistical analyses.

#### **Unscheduled Visits**

- Unscheduled visits will not be included in summary tables.
- Unscheduled visits will not be included in figures.

| Reporting Standard | s |
|---|---|
| All unscheduled visits will be included in listings. | |
| <b>Descriptive Summa</b> | ry Statistics |
| Continuous Data | Refer to IDSL Statistical Principle 6.06.1 |
| Categorical Data | N, n, frequency, % |
| Reporting of Pharm | acokinetic Concentration Data |
| Descriptive | Refer to IDSL Statistical Principle 6.06.1 |
| Summary Statistics | Assign zero to NQ values (Refer to GUI_51487 for further details) |
| Reporting of Pharm | acokinetic Parameters |
| Descriptive<br>Summary Statistics<br>(Log Transformed) | N, n, geometric mean, 95% CI of geometric mean, standard deviation (SD) of logged data and between geometric coefficient of variation (CVb (%)) will be reported. $ \text{CV}_b \text{ (\%)} = \sqrt{\left(\text{exp}(\text{SD}^2) - 1\right) * 100} $ (SD = SD of log transformed data) |
| Parameters Not<br>Being Log<br>Transformed | Tmax |
| Parameters Not<br>Being Summarised | The following PK parameters will not be summarised but listed: %AUCex, Tlast, lambda_z, lambda_z_lower, lambda_z_upper, #pts, R2 |
| Graphical Displays | |
| Refer to IDSL Statistical Principals 7.01 to 7.13. | |

## 10.5. Appendix 5: Derived and Transformed Data

#### 10.5.1. General

## **Multiple Measurements at One Time Point**

- Mean of the measurements will be calculated and used in any derivation of summary statistics but if listed, all data will be presented.
- If there are two values within a time window the value closest to the target day for that window will be used. If values are the same distance from the target then the mean will be taken.
- Subjects having both High and Low values for Normal Ranges at any post-baseline visits for safety parameters will be counted in both the High and Low categories of "Any visit postbaseline" row of related summary tables. This will also be applicable to relevant Potential Clinical Importance summary tables.

#### **Study Day**

- Calculated as the number of days from study day of start of dosing date :
  - Ref Date = Missing
- → Study Day = Missing
- Ref Date < Dosing Start Date → Study Day = Ref Date Dosing Start Date</p>
- Ref Data ≥ Dosing Start Date → Study Day = Ref Date (Dosing Start Date) + 1

## 10.5.2. Study Population

#### **Demographics**

#### Age

- GSK standard IDSL algorithms will be used for calculating age where birth date will be imputed as:
  - Any subject with a missing day will have this imputed as day '15'.
  - Any subject with a missing date and month will have this imputed as '30th June'.
- Birth date will be presented in listings as 'YYYY'.
- Reference date for calculation of age at screening will be from visit 1 (Screening visit) date, however this will be from screen failure date for a screen failure subject.
- Analysis age group will be categorized (Years):
  - <=18, 19-64, 65-74, >=75
- Age will be categorized for EudraCT: Adults (18-64 years)

#### **Body Mass Index (BMI)**

• Calculated as Weight (kg) / [Height (m)<sup>2</sup>

#### 10.5.3. Safety

#### **ECG Parameters**

#### RR Interval

IF RR interval (msec) is not provided directly, then RR can be derived as :

[1] If QTcB is machine read & QTcF is not provided, then :

$$RR = \left[ \left( \frac{QT}{QTcB} \right)^2 \right] * 1000$$

[2] If QTcF is machine read and QTcB is not provided, then:

$$RR = \left[ \left( \frac{QT}{QTeF} \right)^3 \right] * 1000$$

• If ECGs are manually read, the RR value preceding the measurement QT interval should be a collected value THEN do not derive.

#### **Corrected QT Intervals**

- When not entered directly in the eCRF, corrected QT intervals by Bazett's (QTcB) and Fredericia's (QTcF) formulas will be calculated, in msec, depending on the availability of other measurements.
- IF RR interval (msec) is provided then missing QTcB and/or QTcF will be derived as :

$$QTcB = \frac{QT}{\sqrt{\frac{RR}{1000}}}$$

$$QTcF = \frac{QT}{3\sqrt{\frac{RR}{1000}}}$$

#### **Laboratory Parameters**

- If a laboratory value which is expected to have a numeric value for summary purposes, has a non-detectable level reported in the database, where the numeric value is missing, but typically a character value starting with '<x' or '>x' (or indicated as less than x or greater than x in the comment field) is present, the number of significant digits in the observed values will be used to determine how much to add or subtract in order to impute the corresponding numeric value.
  - $\circ$  Example 1: 2 Significant Digits = '< x ' becomes x 0.01
  - Example 2: 1 Significant Digit = '> x' becomes x + 0.1
  - Example 3: 0 Significant Digits = '< x' becomes x 1

| Laboratory Assessments | |
|---|---|
| Haematology | Platelet Count, RBC Count, Haemoglobin, Hematocrit, RBC Indices (MCV, MCH, MCH, %Reticulocytes), WBC count with Differential (Neutrophils, Lymphocytes, Monocytes, Eosinophils, Basophils) |
| Clinical Chemistry | BUN, Creatinine, Glucose (fasting), Potassium, Sodium, Calcium, Aspartate Aminotransferase (AST), Alanine Aminotransferase (ALT), Alkaline phosphatise, Total and direct bilirubin, Total Protein |
| Routine Urinalysis | Specific gravity, pH (assessed by dipstick) • glucose, protein, blood, ketones, bilirubin, urobilinogen, nitrite, leukocyte esterase by dipstick |

#### **Laboratory Assessments**

Microscopic examination (if blood or protein is abnormal)

#### ECG (12-lead ECG)

ECG findings, ECG values (Heart rate, PR interval, QRS duration, QT interval, and QTcF intervals)

#### **Vital Signs**

Pulse rate, Blood pressure (Systolic, Diastolic), respiratory rate, Temperature

#### 10.5.4. Pharmacokinetic

#### **PK Parameters**

- If one or more non-quantifiable (NQ) values occur in a profile before the first measurable
  concentration, they will be assigned a value of zero concentration. For linear plots, zero
  concentration value(s) before the first measurable concentration will be included in the plot. For
  log-linear plots, zero concentration value(s) before the first measurable concentration will be
  assigned a missing value.
- If a single NQ value occurs between measurable concentrations in a profile, the NQ should generally be set to missing in the derivation of pharmacokinetic parameters, statistical analysis, and the individual subject plots.
- If two or more NQ values occur in succession between measurable concentrations, the profile
  will be deemed to have terminated at the last measurable concentration prior to these NQs. For
  the purpose of individual subject plots, these NQs will be set to 0, and the subsequent
  measurable concentrations will be retained. For the derivation of pharmacokinetic parameters,
  these NQs and any subsequent measurable concentrations will be set to missing.
- NQs which occur after the last measurable concentration will be omitted (set to missing) in the
  derivation of pharmacokinetic parameters and from the individual subject plots.
- Individual's PK parameters reported as 'NC' (Not Calculable) or 'ND' (Not Determined) will be
  included in listings but omitted (set to missing) from figures, summaries and statistical analyses.

# 10.6. Appendix 6: Premature Withdrawals & Handling of Missing Data

# 10.6.1. Premature Withdrawals

| Element | Reporting Detail |
|---|---|
| General | Subject study completion was defined as a participant has completed all phases of the study including the last visit or the last scheduled procedure (Follow-up) as described in the protocol. |
| | Withdrawn subjects maybe replaced in the study. |
| | All available data from subjects who were withdrawn from the study will be listed and all available planned data will be included in summary tables and figures, unless otherwise specified. |

# 10.6.2. Handling of Missing Data

| Element | Reporting Detail |
|---|---|
| General | Missing data occurs when any requested data is not provided, leading to blank fields on the collection instrument: |
| | <ul> <li>These data will be indicated by the use of a "blank" in subject listing displays.</li> <li>Unless all data for a specific visit are missing in which case the data is excluded from the table.</li> </ul> |
| | <ul> <li>Answers such as "Not applicable" and "Not evaluable" are not considered to be<br/>missing data and should be displayed as such.</li> </ul> |

# 10.6.2.1. Handling of Partial Dates

| Element | Reporting Detail |
|---|---|
| Concomitant<br>Medications | imputed using the following convention: |
| | <ul> <li>If the partial date is a start date, a '01' will be used for the day and 'Jan' will<br/>be used for the month</li> </ul> |
| | <ul> <li>If the partial date is a stop date, a '28/29/30/31' will be used for the day<br/>(dependent on the month and year) and 'Dec' will be used for the month.</li> </ul> |
| | The recorded partial date will be displayed in listings. |

# 10.7. Appendix 7: Values of Potential Clinical Importance

# 10.7.1. Laboratory Values

| Haematology | | | | |
|---|---|---|---|---|
| <b>Laboratory Parameter</b> | Units | Category | Clinical Concern Range | |
| | | | Low Flag (< x) | High Flag (>x) |
| | | Male | | 0.54 |
| Hematocrit | Ratio of 1 | Female | | 0.54 |
| | | $\Delta$ from BL | ↓0.075 | |
| | /1 | Male | | 180 |
| Hemoglobin | g/L | Female | | 180 |
| | | $\Delta$ from BL | <b>↓25</b> | |
| Lymphocytes | x109/ L | | 8.0 | |
| Neutrophil Count | x109/ L | | 1.5 | |
| Platelet Count | x109/ L | | 100 | 550 |
| While Blood Cell Count (WBC) | x10 <sup>9</sup> / L | | 3 | 20 |

| Clinical Chemistry | | | | |
|---|---|---|---|---|
| Laboratory Parameter | Units | Category | Clinical Concern Range | |
| | | | Low Flag (< x) | High Flag (>x) |
| Calcium | mmol/L | | 2 | 2.75 |
| Creatinine | μmol/L | $\Delta$ from BL | | ↑ 44.2 |
| Glucose | mmol/L | | 3 | 9 |
| Potassium | mmol/L | | 3 | 5.5 |
| Sodium | mmol/L | | 130 | 150 |

| Liver Function | | | |
|--------------------|--------|----------|------------------------|
| Test Analyte | Units | Category | Clinical Concern Range |
| ALT/SGPT | U/L | High | ≥ 2x ULN |
| AST/SGOT | U/L | High | ≥ 2x ULN |
| AlkPhos | U/L | High | ≥ 2x ULN |
| T Bilirubin | µmol/L | High | ≥ 1.5xULN |
| | µmol/L | | 1.5xULN T. Bilirubin |
| T. Bilirubin + ALT | | High | + |
| | U/L | | ≥ 2x ULN ALT |

# 10.7.2. ECG

| ECG Parameter | Units | Clinical Cor | ncern Range |
|----------------------------|-------|--------------|-------------|
| | | Lower | Upper |
| Absolute | | | |
| Absolute QTc Interval | msec | | > 450 [1] |
| Absolute PR Interval | msec | < 110 [1] | > 220 [1] |
| Absolute QRS Interval | msec | < 75 [1] | > 110 [1] |
| Change from Baseline | | | |
| Increase from Baseline QTc | msec | | > 60 [1] |

# NOTES:

# 10.7.3. Vital Signs

| Vital Sign Parameter | Units | Clinical Con | cern Range |
|--------------------------|-------|--------------|------------|
| (Absolute) | | Lower | Upper |
| Systolic Blood Pressure | mmHg | < 85 | > 160 |
| Diastolic Blood Pressure | mmHg | < 45 | > 100 |
| Heart Rate | bpm | < 40 | > 110 |

<sup>1.</sup> Represent standard ECG values of PCI for HV studies

# 10.8. Appendix 8 – Abbreviations & Trade Marks

# 10.8.1. Abbreviations

| Abbreviation | Description |
|---|---|
| ADaM | Analysis Data Model |
| AE | Adverse Event |
| A&R | Analysis and Reporting |
| AUC | Area under the concentration-time curve |
| AUC(0-inf) | Area under the concentration-time curve from time 0 to infinity |
| CDISC | Clinical Data Interchange Standards Consortium |
| CI | Confidence Interval |
| Cmax | Maximum observed concentration |
| CSR | Clinical Study Report |
| $CV_b$ | Coefficient of Variation (Between) |
| eCRF | Electronic Case Record Form |
| ICF | Informed Consent Form |
| ICH | International Conference on Harmonisation |
| IDSL | Integrated Data Standards Library |
| GUI | Guidance |
| PCI | Potential Clinical Importance |
| PDMP | Protocol Deviation Management Plan |
| PK | Pharmacokinetic |
| QTcF | Frederica's QT Interval Corrected for Heart Rate |
| QTcB | Bazett's QT Interval Corrected for Heart Rate |
| RAP | Reporting & Analysis Plan |
| SAC | Statistical Analysis Complete |
| SDTM | Study Data Tabulation Model |
| TFL | Tables, Figures & Listings |
| GSK | GlaxoSmithKline |

# 10.8.2. Trademarks

| Trade | marks of the GlaxoSmithKline<br>Group of Companies |
|-------|----------------------------------------------------|
| NONE | |

| Trademarks not owned by the GlaxoSmithKline Group of Companies |
|----------------------------------------------------------------|
| SAS |
| WinNonlin |

# 10.9. Appendix 9: List of Data Displays

## 10.9.1. Data Display Numbering

The following numbering will be applied for RAP generated displays:

| Section | Tables | Figures |
|------------------|-------------|-------------|
| Study Population | 1.1 to 1.7 | N/A |
| Safety | 2.1 to 2.17 | N/A |
| Pharmacokinetic | 3.1 to 3.3 | 4.1 to 4.13 |
| Section | Listings | |
| ICH Listings | 1 to 36 | |
| Other Listings | N/A | |

### 10.9.2. Mock Example Shell Referencing

Non IDSL specifications will be referenced as indicated and if required an example mock-up displays provided in Appendix 10: Example Mock Shells for Data Displays.

| Section | Figure | Table | Listing |
|------------------|---------|---------|---------|
| Study Population | POP_Fn | POP_Tn | POP_Ln |
| Safety | SAFE_Fn | SAFE_Tn | SAFE_Ln |
| Pharmacokinetic | PK_Fn | PK_Tn | PK_Ln |

#### NOTES:

 Non-Standard displays are indicated in the 'IDSL / TST ID / Example Shell' or 'Programming Notes' column as '[Non-Standard] + Reference.'

# 10.9.3. Deliverable [Priority]

| Delivery [Priority] [1] | Description |
|-------------------------|-------------------------------------|
| SAC [X] | Final Statistical Analysis Complete |

#### NOTES:

1. Indicates priority (i.e. order) in which displays will be generated for the reporting effort.

# 10.9.4. Study Population Tables

| Study F | Study Population Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Subject | Disposition | | | | |
| 1.1. | Safety | ES1 | Summary of Subject Disposition | Completed or withdrawn and the reason for withdrawal. | SAC [1] |
| 1.2. | Screened | ES6 | Summary of Screening Status and Reasons for Screen Failure | The number (%) of Randomized or screening failure subjects as the screening status, and the reason for screening failure. | SAC [1] |
| Protoco | ol Deviation | | | | |
| 1.3. | Safety | DV1 | Summary of Important Protocol Deviations | Data is from DV dataset. | SAC [1] |
| Popula | tion Analysed | | | | |
| 1.4. | Safety | SP1 | Summary of Study Populations | | SAC [1] |
| Demog | Demographic and Baseline Characteristics | | | | |
| 1.5. | Safety | DM1 | Summary of Demographic Characteristics | | SAC [1] |
| 1.6. | Screened | DM11 | Summary of Age Ranges | Adults (18-64 years) | |
| 1.7. | Safety | DM5 | Summary of Race and Racial Combinations | | SAC [1] |

# 10.9.5. Safety Tables

| Safety | : Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Advers | e Events (AEs) | | | | |
| 2.1. | Safety | AE1 | Summary of All Adverse Events by System Organ Class and Preferred Term | | SAC [1] |
| 2.2. | Safety | AE5A | Summary of All Adverse Events by Maximum Intensity | | SAC [1] |
| 2.3. | Safety | AE1 | Summary of All Drug-Related Adverse Events by System Organ Class and Preferred Term | | SAC [1] |
| 2.4. | Safety | AE5A | Summary of All Drug-Related Adverse Events by Maximum Intensity | | SAC [1] |
| Labora | tory: Chemistry | y | | | |
| 2.5. | Safety | LB1 | Summary of Chemistry | | SAC [1] |
| 2.6. | Safety | LB1 | Summary of Chemistry Changes from Baseline | | SAC [1] |
| 2.7. | Safety | LB4 | Summary of Chemistry Data Shifts from Baseline with Respect to the Normal Range | | SAC [1] |
| Labora | tory: Hematolo | gy | | | |
| 2.8. | Safety | LB1 | Summary of Hematology | | SAC [1] |
| 2.9. | Safety | LB1 | Summary of Hematology Changes from Baseline | | SAC [1] |
| 2.10. | Safety | LB4 | Summary of Hematology Data Shifts from Baseline with Respect to the Normal Range | | SAC [1] |

| Safety | Safety : Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Labora | tory: Urinalysis | <b>,</b> | | | |
| 2.11. | Safety | UR3b | Summary of Urinalysis (Glucose, Protein, Blood, Ketones, Bilirubin, Urobilinogen nitrite, leukocyte esterase) Data | | SAC [1] |
| 2.12. | Safety | LB1 | Summary of Urinalysis (Specific Gravity and pH) | | SAC [1] |
| ECG | | | | | |
| 2.13. | Safety | EG1 | Summary of ECG Findings | | SAC [1] |
| 2.14. | Safety | EG2 | Summary of ECG Value | | SAC [1] |
| 2.15. | Safety | EG2 | Summary of Change from Baseline in ECG Values by Visit | | SAC [1] |
| Vital Si | Vital Signs | | | | |
| 2.16. | Safety | VS1 | Summary of Vital Signs | | SAC [1] |
| 2.17. | Safety | VS1 | Summary of Change from Baseline in Vital Signs | | SAC [1] |

# 10.9.6. Pharmacokinetic Tables

| Pharma | Pharmacokinetic : Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.1. | PK | PK01: PKCT1 | Summary of Pyrimethamine Plasma Concentration | | SAC [1] |
| 3.2. | PK | PK03: PKPT1 | Summary of Pyrimethamine Pharmacokinetic Parameters (non-transformed) | | SAC [1] |
| 3.3. | PK | PK05: PKPT3 | Summary of Pyrimethamine Pharmacokinetic Parameters (loge-transformed) | | SAC [1] |

# 10.9.7. Pharmacokinetic Figures

| Pharmacokinetic: Figures | | | | | |
|---|---|---|---|---|---|
| IDSL /<br>TST<br>ID /<br>Exam<br>ple<br>Shell | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 4.1. | PK | PK16a:<br>PKCF1p | Individual Pyrimethamine Plasma Concentration-Time Plots by Subject (from Pre-Dose to Day 22) | by Subject (Linear and Semi-Log) Time: from Pre-dose to Day 22 | SAC [1] |
| 4.2. | PK | PK24: pkcf6 | Individual Pyrimethamine Plasma Concentration-Time Plots by group (from Pre Dose to Day 22) | By group (Linear and Semi-Log) Time: from Pre-dose to Day 22 | SAC [1] |
| 4.3. | PK | PK19: PKCF4 | Mean (+SD) Pyrimethamine Concentration-Time Plots (from Pre Dose to Day 22) | Time: from Pre-dose to Day 22 | SAC [1] |
| 4.4. | PK | PK18: PKCF3 | Median Pyrimethamine Plasma Concentration-Time Plots (from Pre Dose to Day 22) | Time: from Pre-dose to Day 22 | SAC [1] |
| 4.5. | PK | PK16a:<br>PKCF1p | Individual Pyrimethamine Plasma Concentration-Time Plots by Subject (from Pre Dose to 72 hr) | by Subject (Linear and Semi-Log) Time: from Pre-dose to 72 hr | SAC [1] |
| 4.6. | PK | PK24: pkcf6 | Individual Pyrimethamine Plasma Concentration-Time Plots by group (from Pre Dose to 72 hr) | By rgroup (Linear and Semi-Log) Time: from Pre-dose to 72 hr | SAC [1] |
| 4.7. | PK | PK19: PKCF4 | Mean (+SD) Pyrimethamine Concentration-Time Plots (from Pre Dose to 72 hr) | Time: from Pre-dose to 72 hr | SAC [1] |
| 4.8. | PK | PK18: PKCF3 | Median Pyrimethamine Plasma Concentration-Time Plots (from Pre Dose to 72 hr) | Time: from Pre-dose to 72 hr | SAC [1] |
| 4.9. | PK | PK28 | Plot of Pyrimethamine Treatment and PK Parameters | AUC(0-t), AUC(0-inf), Cmax, t1/2 Plot and Mean with 95%CI X axis: Japanese, Caucasian Y axis: PK parameters | SAC [1] |

| Pharma | Pharmacokinetic: Figures | | | | |
|---|---|---|---|---|---|
| IDSL /<br>TST<br>ID /<br>Exam<br>ple<br>Shell | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 4.10. | PK | Study Specifics<br>(PK_F1) | Individual Pyrimethamine Plasma Concentration-Time Plots (from Pre-Dose to Day 22) | Japanese & Caucasian<br>(Linear and Semi-Log)<br>Time: from Pre-dose to Day 22 | SAC [1] |
| 4.11. | PK | Study Specifics<br>(PK_F1) | Individual Pyrimethamine Plasma Concentration-Time Plots (from Pre-Dose to 72 hr) | Japanese & Caucasian<br>(Linear and Semi-Log)<br>Time: from Pre-dose to 72 hr | SAC [1] |
| 4.12. | PK | Study Specifics<br>(PK_F2) | Mean (+SD) Pyrimethamine Concentration-Time Plots (from Pre Dose to Day 22) | Japanese & Caucasian<br>Time: from Pre-dose to Day 22 | SAC [1] |
| 4.13. | PK | Study Specifics (PK_F2) | Mean (+SD) Pyrimethamine Concentration-Time Plots (from Pre Dose to 72 hr) | Japanese & Caucasian<br>Time: from Pre-dose to 72 hr | SAC [1] |

# 10.9.8. ICH Listings

Note: 'Inv.' in the standard displays will be replaced to 'Centre'.

| ICH : L | ICH : Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Subjec | Subject Disposition | | | | |
| 1. | Screening<br>Failure | ES7 | Listing of Reasons for Screen Failure | | SAC [1] |
| 2. | Safety | ES2 | Listing of Reasons for Study Withdrawal | | SAC [1] |
| Protoc | ol Deviations | | | | |
| 3. | Safety | DV2 | Listing of Important Protocol Deviations | | SAC [1] |
| 4. | Screened | IE4 | Listing of Subjects with Inclusion/Exclusion Criteria Deviations | | SAC [1] |
| Popula | tions Analysed | | | | |
| 5. | Safety | Study Specifics (SP_T1) | Listing of Subjects Excluded from PK Population | | SAC [1] |
| Demog | raphic and Bas | eline Characteris | tics | | |
| 6. | Safety | DM2 | Listing of Demographic Characteristics | "Age at Screening" is added. | SAC [1] |
| 7. | Screening<br>Failure | DM2 | Listing of Demographic Characteristics for Screening Failure Subjects | | SAC [1] |
| 8. | Safety | DM9 | Listing of Race | | SAC [1] |
| 9. | Screening<br>Failure | DM9 | Listing of Race for Screening Failure Subjects | | SAC [1] |
| Medica | Medical Conditions and Concomitant Medications | | | | |
| 10. | Screened | MH3 | Listing of Medical Conditions | | SAC [1] |

| ICH : Listings | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 11. | Safety | CM5 | Listing of Concomitant Medications | | SAC [1] |
| 12. | Safety | CM6 | Relationship between ATC Level 1, Ingredient and Verbatim Text | | SAC [1] |
| Exposi | ire and Treatmo | ent Compliance | | | |
| 13. | Safety | EX3 | Listing of Exposure Data | | SAC [1] |
| Advers | e Events | | | | |
| 14. | Safety | CP_AE8 | Listing of All Adverse Events | | SAC [1] |
| 15. | Safety | AE7 | Listing of Subject Numbers for Individual Adverse Events | | SAC [1] |
| 16. | Screened | AE2 | Listing of Relationship Between Adverse Event System Organ Classes, Preferred Terms, and Verbatim Text | | SAC [1] |
| Serious | Serious and Other Significant Adverse Events | | | | |
| 17. | Safety | CP_AE8 | Listing of Serious Adverse Events | | SAC [1] |
| 18. | Screening<br>Failure | CP_AE8 | Listing of Serious Adverse Events for Screening Failure Subject | | SAC [1] |
| 19. | Safety | CP_AE8 | Listing of Adverse Events Leading to Withdrawal from Study | | SAC [1] |
| Labora | tory (Chemistry | / Data) | | | |
| 20. | Safety | CP_LB5 | Listing of All Chemistry Data | Change from baseline is included. | SAC [1] |
| 21. | Safety | CP_LB5 | Listing of All Chemistry Data for Subjects with Any Value of Potential Clinical Importance | | SAC [1] |
| Labora | tory (Hematolo | gy Data) | | | |
| 22. | Safety | CP_LB5 | Listing of All Hematology Data | Change from baseline is included. | SAC [1] |
| 23. | Safety | CP_LB5 | Listing of All Hematology Data for Subjects with Any Value of Potential Clinical Importance | | SAC [1] |

| ICH : Listings | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Labora | Laboratory (Urinalysis Data) | | | | |
| 24. | Safety | UR2a | Listing of All Urinalysis Dipstick and Microscopy Data | Time will be displayed after 'Date'. | SAC [1] |
| 25. | Safety | CP_LB5 | Listing of Urinalysis Data (Gravity and pH) | | SAC [1] |
| Hepato | biliary (Liver) | | | | |
| 26. | Safety | LIVER5 | Listing of Liver Monitoring/Stopping Event Reporting | | SAC [1] |
| 27. | Safety | MH2 | Listing of Medical Conditions for Subjects with Liver Stopping<br>Events | | SAC [1] |
| 28. | Safety | SU2 | Listing of Substance Use for Subjects with Liver Stopping Events | | SAC [1] |
| ECG | | | | | |
| 29. | Safety | EG3 | Listing of All ECG Values | | SAC [1] |
| 30. | Safety | EG3 | Listing of Change from Baseline in ECG Values | | SAC [1] |
| 31. | Safety | EG5 | Listing of ECG Findings | | SAC [1] |
| 32. | Safety | CP_EG3 | Listing of All ECG Data for Subjects with Any Value of Potential Clinical Importance | | SAC [1] |
| Vital Si | gns | | | | |
| 33. | Safety | VS4 | Listing of All Vital Signs | Change from baseline is included. | SAC [1] |
| 34. | Safety | CP_VS4 | Listing of All Vital Signs Data for Subjects with Any Value of Potential Clinical Importance | | SAC [1] |
| PK | | | | | |
| 35. | PK | PK07: PKCL1p | Listing of Pyrimethamine Plasma Concentration | | SAC [1] |
| 36. | PK | PK13: PKPL1p | Listing of Pyrimethamine Pharmacokinetic Parameters | | SAC [1] |

# 10.10. Appendix 10: Example Mock Shells for Data Displays

Example: PK\_F1
Protocol: 12345
Page 1 of 1

Population: PK

Table X
Individual Plasma Concentration-Time Plots



NOTE: LLQ = XX unit

USER ID:directory/program.sas 27JUN2014 12:00

Example: PK\_F2
Protocol: 12345

Protocol: 12345
Population: PK

Table X

Mean + SD Concentration-Time Plots (Linear and Semi-log)



NOTE: LLQ = XX unit
USER ID:directory/program.sas 27JUN2014 12:00